CLINICAL TRIAL: NCT03645837
Title: Reducing Compression Duration Post Trans Radial Cardiac Catheterization
Brief Title: Rapid Clamp Release Post Trans-radial Cardiac Catheterization
Acronym: PRACTICAL-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112619
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Catheterization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10 minutes (Experimental): Compression clamp release start after 10 minutes
  Interventions: Other: Compression clamp release
- 20 minutes (Experimental): Compression clamp release start after 20 minutes
  Interventions: Other: Compression clamp release
- 30 minutes (Active Comparator): Compression clamp release start after 30 minutes
  Interventions: Other: Compression clamp release

INTERVENTIONS:
Other: Compression clamp release — Standard compression clamp is used and will be released at different times according to randomization

SUMMARY:
The purpose of the study is to compare different short durations of radial clamp application following an angiogram via a trans-radial approach.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized study that will enroll patients that are referred for an angiogram and will compare 3 different durations of radial clamp applications. Patients will be randomly assigned to either 10, 20 or 30-minute clamp applications. The clamps will be gradually released at the end of the assigned durations and participants will be assessed for the radial artery occlusion, hematoma, and other bleeding events.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic catheterization
2. 5 F slender sheath
3. Normal ulno-palmar circulation

Exclusion Criteria:

1. Abnormal ulno-palmar circulation type D
2. Ad hoc percutaneous coronary intervention
3. Heparin or other anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Hematoma | 1 hour
  Hematoma larger than 5 cm
Radial artery occlusion | 1 hour
  Assessed by Doppler

SECONDARY OUTCOMES:
Bleeding - any | 1 hour
  Minor hematoma

OTHER OUTCOMES:
Comparison to prior study results | 1 hour
  Compared to PRACTICAL study

CONTACTS AND LOCATIONS:
Overall Officials: Shahar Lavi, MD, Principal Investigator — London Health Sceinces Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavi S, Cheema A, Yadegari A, Israeli Z, Levi Y, Wall S, Alemayehu M, Parviz Y, Murariu BD, McPherson T, Syed J, Bagur R. Randomized Trial of Compression Duration After Transradial Cardiac Catheterization and Intervention. J Am Heart Assoc. 2017 Feb 3;6(2):e005029. doi: 10.1161/JAHA.116.005029. PMID 28159821